CLINICAL TRIAL: NCT05298709
Title: Functional Magnetic Resonance Imaging (fMRI) Vascular Reactivity in Cerebral Cavernous Malformations (CCM)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was determined to not be feasible at this time.
Sponsor: University of New Mexico (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-136
Record Dates: First submitted 2022-03-09; First posted 2022-03-28 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cerebral Cavernous Malformation
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypercarbia/Hypocarbia/resting state during fMRI (Experimental): During real time fMRI, all subjects will completed breathing tasks though a mask that supplies gas mixtures using the RespirAct™ Gas Control System (Thornhill Medical). The RespirAct™ is a computer-controlled gas blender providing carbon dioxide (CO2), oxygen (O2) and nitrogen for a subject to inhale while breathing for the purpose of controlling the concentrations of the respective blood gases.
  For hypocarbia, subjects will be instructed to pace their breathing to 16- 20 breaths-per-minute to achieve a stable target end-tidal CO2 between 30 and 40 mm Hg.
  Hypercarbia will be induced by increasing CO2 concentration and flow rate of the gas mixture until a desired ETCO2 level between 40 and 50 mm Hg has been reached.
  There will also be a 10 minutes rest period during which respiratory rate and heart rate will be monitored continuously.
  Interventions: Other: Hyperventilation and CO2 challenge

INTERVENTIONS:
Other: Hyperventilation and CO2 challenge — Subjects will also be asked to complete hyperventilation and CO2 breathing tasks based on instruction from the study investigators as described in study arm.

SUMMARY:
The goal is to characterize vascular reactivity and cardiac pulsatility of normal appearing white matter in patients with CCM during hypercarbia/hypocarbia using quantitative real-time high-speed multi-echo fMRI to develop prognostic biomarkers for CCM formation

ELIGIBILITY:
Inclusion Criteria:

1. All familial CCM subjects presenting at UNMH who can consent to our study.
2. Adult Male/Female patients ages >18 years old

Exclusion Criteria:

1. Individuals ages <18 year
2. Subjects with a known fear of dyspnea or enclosed spaces will be excluded from this study as well as those with metal implants, COPD, heart conditions, and hypercapnia.
3. Subjects who have contraindications to MRI such as harboring incompatible ferromagnetic objects implanted in the body.
4. Pregnant women (screening for pregnancy will be performed by oral questionnaire. MRI is safe in pregnancy but the study will exclude pregnant subjects, as the effects of respiratory challenge cannot be predicted in such subjects. Since these effects are proportional to the stage of gestation, oral history will be sufficient to assure safety.)
5. Prisoners.
6. People unable to consent.
7. People unable to participate due to prior neurological deficits.
8. Subjects with underlying pre-existing pulmonary illness; such as asthma, COPD, pulmonary hypertension, will be excluded.
9. Cognitively impaired and/or participants not able to speak English language will not be included in the study (This pilot study involves performing motor and verbal tasks while in the MRI, in addition to undergoing a respiratory challenge, that requires understanding instructions clearly. We do not have current capabilities to include a translator who would be available at all stages of the study to include subjects who do not speak English.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-07-17 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Response | 12 Months
  Primary end point of the study is to measure the amplitude and frequency response of hemodynamic response function during hypercarbia/hypocarbia using task-based functional MRI
Resting state connectivity | 12 month
  To measure the strength of resting-state connectivity during hypercarbia/hypocarbia using high-speed multi-echo resting-state functional MRI.

SECONDARY OUTCOMES:
Cardiac Pulsatility | 12 Months
  Measure the amplitude and frequency spectrum of the cardiac pulsatility during hypercarbia/hypocarbia in functional MRI time series that are acquired using high-speed multi-echo functional MRI
First Harmonic | 12 Months
  To measure the amplitude ratio of the first harmonic of the cardiac pulsatility relative to the cardiac base frequency in these data, which is a biomarker of vascular compliance.speed multi echo fMRI.

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Neurology Research Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
There would not be any plans in place to share IPD. All data will be de-identified and not linked to any individual participant.